CLINICAL TRIAL: NCT06783023
Title: Evaluation of the Validity and Reliability of the '6 Minute Pegboard and Ring Test' Unsupported Arm Function Exercise Test in Patients Using Pacemakers
Status: Recruiting | Type: Observational
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gamze Nur AHISKALI, Physiotherapist Gamze Nur AHISKALI, Erol Olcok Corum Training and Research Hospital
Other Study IDs: 2024-08/2
Record Dates: First submitted 2024-09-10; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Implantable Electrical Devices; Upper Extremity Function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Implantable Electronic Devices: individuals with cardiac implantable electronic devices
  Interventions: Other: validity and reliability study

INTERVENTIONS:
Other: validity and reliability study — In the study, which will include at least 24 individuals with CIED determined by power analysis, unassisted arm exercise capacity and arm function/endurance, maximum arm exercise capacity, double product, heart recovery, comorbidity level, hand grip strength, fear of movement, activities of daily living and quality of life will be evaluated.

SUMMARY:
Recently, the use of Cardiac Implantable Electronic Devices (CIED) is becoming widespread due to the improvement of patients' symptoms, reduction of sudden cardiac death and improved quality of life. Although implantation of the device is considered a minor invasive procedure, possible but often underestimated dysfunction of the same side upper extremity may develop after implantation. This increase in the number of device implantations makes shoulder dysfunction after pacemaker implantation a major health problem. In the current research in the literature, arm dysfunction is evaluated by measuring range of motion with a dynamic goniometer, scales scored independently of shoulder pathology and the effect of activities of daily living. This indicates that there is no objective functional assessment method used to evaluate arm function in CIED patients. Therefore, the point of this study is to find out how reliable and valid the 6 Minute Pegboard and Ring Test (6PBRT) is for testing the functional capacity of the upper extremity in people who have had CIED implanted.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65 who have a pacemaker,
* At least 3 months have passed since pacemaker implantation and there are no complications in the last pacemaker control,
* Being in NYHA class I-II-III,
* Patients with no coordination problems,
* Patients who volunteered to participate in the study.

Exclusion Criteria:

* Patients with a history of shoulder pathologies prior to pacemaker implantation that may restrict movement of the upper limb (conditions such as severe pain around the shoulder, edema or shoulder dislocation that may restrict upper limb movement),
* Patients with a history of shoulder surgery (limitation in range of motion),
* Patients who have had a cerebrovascular event resulting in mastectomy or arm involvement on the affected side,
* Patients with decompensated heart failure,
* Patients with a history of ICD inappropriate shock,
* Those with acute myocardial infarction,
* Patients with malignancy on active treatment, collagen tissue disease receiving systemic steroids,
* Chronic kidney disease patients on dialysis with unstable volume load.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with implantable cardiac electrical devices
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of unsupported arm exercise capacity | 1 year
  6 Minute Pegboard and Ring Test-6PBRT
Evaluation of maximal arm exercise capacity | 1 year
  Arm Ergometer Test / It is a gold standard method used to evaluate upper extremity exercise capacity. At the beginning and end of the test, heart rate, saturation and BORG scale will be evaluated for fatigue and dyspnea. In women, it will start with 20 watts and increase by 6 watts every 1 minute, while in men, it will start with 30 watts and increase by 10 watts every 1 minute. The rotation speed will be maintained at 70 rpm. The test will be terminated if the perceived exertion level is ≥ 18 and/or the rotation speed cannot be maintained above 60 rpm.

SECONDARY OUTCOMES:
Evaluation of hand grip strength | 1 year
  JAMAR Hydraulic Hand Dynamometer
Evaluation of Activities of Daily Living | 1 year
  Performance Measure for Activities of Daily Living-8 for Patient with Mild Symptomatic Heart Failure- PMADL-8. The total score ranges from 8-32, with a high score indicating a level of limitation in activities of daily living.
Evaluation of Quality of Life | 1 year
  MacNew Heart Disease Health-Related Quality of Life Questionnaire / The questions are scored from 1 to 7, with higher scores indicating better quality of life.
Evaluation of Kinesiophobia | 1 year
  Tampa Scale of Kinesiophobia for Heart- TSK- HEART / The person receives a total score between 17 and 68. A high score on the scale indicates a high level of kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Corum Erol Olçok Training and Research Hospital, Çorum, Center, Turkey (Türkiye)